CLINICAL TRIAL: NCT02706873
Title: A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) Once Daily Monotherapy to Methotrexate (MTX) Monotherapy in MTX-Naïve Subjects With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: A Study to Compare Upadacitinib (ABT-494) Monotherapy to Methotrexate (MTX) Monotherapy in Adults With Rheumatoid Arthritis (RA) Who Have Not Previously Taken Methotrexate
Acronym: SELECT-EARLY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-545; 2015-003334-27 (EudraCT Number)
Record Dates: First submitted 2016-02-18; First posted 2016-03-11 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal disease; Arthritis; Joint disease; Anti-inflammatory agents; Antirheumatic agents; ABT-494; Upadacitinib
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — Methotrexate; upadacitinib

STUDY DESIGN:
Intervention Model Description: Participants were to be randomized in a 1:1:1 ratio to treatment Groups 2, 3, and 4 below, except for participants from Japan, who were to be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3, and 4:
  Group 1: Upadacitinib 7.5 mg QD monotherapy (Japan only)
  Group 2: Upadacitinib 15 mg QD monotherapy (43 countries, including Japan)
  Group 3: Upadacitinib 30 mg QD monotherapy (43 countries, including Japan)
  Group 4: MTX monotherapy (43 countries, including Japan)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Methotrexate (Active Comparator): Period 1: Participants will receive placebo to upadacitinib once daily and methotrexate once weekly for 48 weeks.
  Period 2: Participants will continue on placebo to upadacitinib once daily and methotrexate once weekly until the study is unblinded, after which participants will receive open-label methotrexate up to Week 260.
  Interventions: Drug: Placebo to Upadacitinib; Drug: Methotrexate
- Upadacitinib 7.5 mg (Japan-only) (Experimental): Period 1: Participants will receive upadacitinib 7.5 mg once daily and placebo to methotrexate once weekly for 48 weeks.
  Period 2: Participants will continue on upadacitinib 7.5 mg once daily and placebo to methotrexate once weekly until the study is unblinded, after which participants will receive open-label upadacitinib 7.5 mg up to Week 260.
  Interventions: Drug: Placebo to Methotrexate; Drug: Upadacitinib
- Upadacitinib 15 mg (Experimental): Period 1: Participants will receive upadacitinib 15 mg once daily and placebo to methotrexate once weekly for 48 weeks.
  Period 2: Participants will continue on upadacitinib 15 mg once daily and placebo to methotrexate once weekly until the study is unblinded, after which participants will receive open-label upadacitinib 15 mg up to Week 260.
  Interventions: Drug: Placebo to Methotrexate; Drug: Upadacitinib
- Upadacitinib 30 mg (Experimental): Period 1: Participants will receive upadacitinib 30 mg once daily and placebo to methotrexate once weekly for 48 weeks.
  Period 2: Participants will continue on upadacitinib 30 mg once daily and placebo to methotrexate once weekly until the study is unblinded, after which participants will receive open-label upadacitinib 30 mg once daily. After implementation of Protocol Amendment 6 participants will receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Placebo to Methotrexate; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo to Upadacitinib — Tablet; Oral
  Arms: Methotrexate
Drug: Methotrexate — Capsule or Tablet; Oral
  Arms: Methotrexate
Drug: Placebo to Methotrexate — Capsule or Tablet; Oral
  Arms: Upadacitinib 15 mg; Upadacitinib 30 mg; Upadacitinib 7.5 mg (Japan-only)
Drug: Upadacitinib — Tablet; Oral
  Other Names: ABT-494; Rinvoq
  Arms: Upadacitinib 15 mg; Upadacitinib 30 mg; Upadacitinib 7.5 mg (Japan-only)

SUMMARY:
The objectives of Period 1 were the following:

* To compare the safety and efficacy of upadacitinib 7.5 mg once daily (QD) monotherapy (for participants in Japan only), 15 mg QD monotherapy, and 30 mg QD monotherapy versus weekly methotrexate monotherapy for the treatment of signs and symptoms of RA in methotrexate-naïve adults with moderately to severely active RA;
* To compare the efficacy of upadacitinib 15 mg QD monotherapy and upadacitinib 30 mg QD monotherapy versus weekly methotrexate monotherapy for prevention of structural progression in methotrexate-naïve adults with moderately to severely active RA.

The objective of Period 2 is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 7.5 mg QD (for participants in Japan only), 15 mg QD, and 30 mg QD in adults with RA who have completed Period 1.

DETAILED DESCRIPTION:
This study includes 2 periods (a 48-week double-blind treatment period and a long-term extension period) and a Japan substudy. In Period 1 participants will be randomized in a 1:1:1 ratio to treatment Groups 2, 3, and 4 below, except for participants from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3, and 4:

* Group 1: Upadacitinib 7.5 mg once daily (QD) monotherapy (participants in Japan only)
* Group 2: Upadacitinib 15 mg QD monotherapy
* Group 3: Upadacitinib 30 mg QD monotherapy
* Group 4: Methotrexate monotherapy

Rescue therapy is defined for Weeks 12 through 24, Week 26, and Weeks 36 through 40. Starting at Week 12 through Week 24, participants who do not achieve ≥ 20% improvement in both tender joint count (TJC) and swollen joint count (SJC) compared with baseline at two consecutive visits will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: non-steroidal anti-inflammatory drug(s) (NSAIDs), corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days) and/or low-potency analgesics.

Rescue therapy for participants who meet the following criteria at Week 26 are as follows:

Participants who do not achieve clinical remission (CR) based on Clinical Disease Activity Index (CDAI) (defined as a CDAI score ≤ 2.8):

* but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded study drug and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low-potency analgesics and conventional synthetic disease-modifying anti-rheumatic drug(s) (csDMARDs) (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
* and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline and originally assigned to methotrexate will be re-randomized in a 1:1 ratio to receive blinded upadacitinib 15 mg QD or upadacitinib 30 mg QD (participants in Japan will be randomized 1:1:1 to receive upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD) while continuing methotrexate treatment in a blinded manner until the study is unblinded. Participants originally assigned to upadacitinib will add methotrexate 10 mg/week (7.5 mg for Japan) to upadacitinib in a blinded manner and will remain on upadacitinib plus methotrexate 10 mg/week (7.5 mg for Japan) until the study is unblinded.

Starting at Week 36 through Week 40, participants who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine).

Participants who complete the Week 48 visit (end of Period 1) will enter the long-term extension, Period 2 (212 weeks) and continue study treatment per assignment at the end of Period 1 in a blinded fashion. When the last participant completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded, and participants will be dispensed study drug in an open-label fashion until the completion of Period 2. Starting with Protocol Amendment 6, participants receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD, and participants receiving methotrexate will receive open-label methotrexate.

A global analysis will be conducted for the comparisons of the primary and secondary efficacy endpoints between the upadacitinib 15 mg QD and 30 mg QD treatment groups versus the methotrexate treatment group for all participants (excluding the Japan specific upadacitinib 7.5 mg treatment group). Analyses will be conducted separately for United States (US)/Food and Drug Administration (FDA), European Union (EU)/European Medicines Agency (EMA), and Japan/Pharmaceuticals and Medical Devices Agency (PMDA) regulatory purposes, each according to a pre-specified sequence of primary and ranked secondary endpoints.

A separate Japan sub-study analysis will be conducted for the comparisons of the efficacy endpoints between the upadacitinib 7.5 mg QD, 15 mg QD, and 30 mg QD treatment groups versus the methotrexate treatment group for participants enrolled in Japan only.

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms consistent with RA for ≥ 6 weeks who also fulfill the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA.
* Naïve to Methotrexate (MTX) or, if already on MTX, have received no more than 3 weekly MTX doses with requirement to complete a 4-week MTX washout before the first dose of study drug.
* Participants with prior exposure to conventional synthetic disease-modifying anti-rheumatic drugs(csDMARDs) other than MTX may be enrolled if completed the washout period.
* Participant meets both of the following minimum disease activity criteria:

  -≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
* high sensitivity C reactive protein (hsCRP) ≥ 5 mg/L (central lab, upper limit of normal [ULN] 2.87 mg/L at Screening Visit.
* Greater than or equal to 1 bone erosion on x-ray (by local reading) OR in the absence of documented bone erosion, both positive rheumatoid factor (RF) and positive anti-cyclic citrullinated peptide (anti CCP) autoantibodies are required at Screening.
* Stable dose of non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, oral corticosteroids (equivalent to prednisone ≤ 10 mg/day), or inhaled corticosteroids for stable medical conditions are allowed but must have been at a stable dose ≥ 1 week prior to the first dose of study drug.

Exclusion Criteria:

* Intolerant to Methotrexate (MTX).
* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Prior exposure to any biologic disease-modifying anti-rheumatic drugs (bDMARDs).
* History of any arthritis with onset prior to age 17 years or current diagnosis, inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [currently with active symptoms]. Current diagnosis of secondary Sjogren's Syndrome is permitted.
* Has been treated with intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, or intra-tendon sheath corticosteroids in the preceding 8 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (290):
- United States (32):
  - TriWest Research Associates- La Mesa /ID# 143738, La Mesa, California
  - Desert Medical Advances /ID# 143730, Palm Desert, California
  - International Medical Research - Daytona /ID# 143748, Daytona Beach, Florida
  - FL Med Ctr and Research, Inc. /ID# 143724, Miami, Florida
  - Millennium Research /ID# 143736, Ormond Beach, Florida
  - Arthritis Research of Florida /ID# 143743, Palm Harbor, Florida
  - Sarasota Arthritis Center /ID# 145978, Sarasota, Florida
  - FL Med Clinic, PA /ID# 143744, Zephyrhills, Florida
  - Deerbrook Medical Associates /ID# 143728, Vernon Hills, Illinois
  - Four Rivers Clinical Research /ID# 143741, Paducah, Kentucky
  - Ocean Rheumatology, PA /ID# 143737, Toms River, New Jersey
  - Arthritis Rheumatic Back Disorder /ID# 143733, Voorhees Township, New Jersey
  - Trinity Health Med Arts Clinic /ID# 143727, Minot, North Dakota
  - STAT Research, Inc. /ID# 143750, Vandalia, Ohio
  - Healthcare Research Consultant /ID# 143747, Tulsa, Oklahoma
  - Advanced Rheumatology & Arthri /ID# 147947, Wexford, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 145653, Summerville, South Carolina
  - West Tennessee Research Inst /ID# 143723, Jackson, Tennessee
  - Dr. Ramesh Gupta /ID# 143732, Memphis, Tennessee
  - Diagnostic Group Integrated He /ID# 152921, Beaumont, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 147626, Corpus Christi, Texas
  - Doctor's Hosp at Renaissance /ID# 156407, Edinburg, Texas
  - MedResearch Inc. /ID# 156409, El Paso, Texas
  - Rheumatic Disease Clin Res Ctr /ID# 151103, Houston, Texas
  - Accurate Clinical Research /ID# 143749, Houston, Texas
  - SW Rheumatology Res. LLC /ID# 143745, Mesquite, Texas
  - Sun Research Institute /ID# 159546, San Antonio, Texas
  - Accurate Clinical Management /ID# 159543, San Antonio, Texas
  - NextGen Clinical Trials LLP /ID# 150930, San Antonio, Texas
  - Arthritis Clinic of Central TX /ID# 159541, San Marcos, Texas
  - Arthritis & Osteoporosis Clinic /ID# 159542, Waco, Texas
  - Arthritis Clinic of N. VA, P.C /ID# 143734, Arlington, Virginia
- Argentina (7):
  - Aprillus Asistencia e Investig /ID# 149179, Capital Federal, Buenos Aires
  - Iari /Id# 148595, San Isidro, Buenos Aires
  - Instituto CAICI /ID# 143141, Rosario, Santa Fe Province
  - Org Medica de Investigacion /ID# 143142, Buenos Aires
  - Consultora Integral de Salud S /ID# 143144, Córdoba
  - Centro Integral de Reumatologi /ID# 143143, San Miguel de Tucumán
  - Centro Medico Privado/Reuma /ID# 143140, San Miguel de Tucumán
- Australia (5):
  - Royal Prince Alfred Hospital /ID# 143149, Camperdown, New South Wales
  - Rheumatology Research Unit /ID# 143147, Maroochydore, Queensland
  - The Queen Elizabeth Hospital /ID# 143148, Woodville, South Australia
  - Southern Clinical Research Pty /ID# 143150, Hobart, Tasmania
  - Emeritus Research /ID# 143146, Camberwell, Victoria
- Belarus (2):
  - First City Clinical Hospital /ID# 159020, Minsk
  - City Clinical Hospital #9 /ID# 145650, Minsk
- Belgium (5):
  - Rhumaconsult SPRL /ID# 143158, Charleroi, Hainaut
  - Algemeen Stedelijk Ziekenhuis /ID# 153504, Aalst, Oost-Vlaanderen
  - UZ Gent /ID# 143157, Ghent, Oost-Vlaanderen
  - ReumaClinic Genk /ID# 143159, Genk
  - CHU Ambroise Pare /ID# 152955, Mons
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic of Srpska /ID# 143161, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 143162, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 143164, Sarajevo
- Brazil (6):
  - CIP - Centro Internacional de Pesquisa /ID# 143171, Goiânia, Goiás
  - Ceti - Centro de Estudos Em Terapias Inovadoras Ltda /Id# 143169, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 143168, Porto Alegre, Rio Grande do Sul
  - LMK Sevicos Medicos S/S /ID# 143167, Porto Alegre, Rio Grande do Sul
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda /ID# 143166, São Paulo, São Paulo
  - CCBR Brasil /ID# 150925, Rio de Janeiro
- Bulgaria (5):
  - MHAT Trimontsium /ID# 143173, Plovdiv
  - UMHAT Pulmed OOD /ID# 143176, Plovdiv
  - MHAT Kaspela /ID# 143172, Plovdiv
  - Diagnostic Consultative Center /ID# 143174, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 143175, Sofia
- Canada (5):
  - Rheumatology Research Assoc /ID# 143206, Edmonton, Alberta
  - Manitoba Clinic /ID# 143203, Winnipeg, Manitoba
  - Ciads /Id# 143205, Winnipeg, Manitoba
  - CA Ctr for Clin Trials CCCT /ID# 159080, Thornhill, Ontario
  - Ctr. de Rheum de l'est du QC /ID# 151317, Rimouski, Quebec
- Chile (7):
  - Ctr de Inv Clinica del Sur /ID# 143208, Temuco, Región de la Araucanía
  - Someal /Id# 143207, Providencia, Santiago Metropolitan
  - Quantum Research LTDA. /ID# 143210, Puerto Varas
  - Quantum Research Stgo. /ID# 145651, Santiago
  - Soc. de Prestaciones medicas y Paramedicas Goecke /ID# 143209, Santiago
  - Investigaciones Medicas SSMSO /ID# 151685, Santiago
  - Centro de Estudios Clinicos Qu /ID# 152913, Viña del Mar
- China (3):
  - 1st Aff Hosp of Bengbu Med Col /ID# 162974, Bengbu, Anhui
  - The 1st Aff Hosp Xiamen Univ /ID# 162076, Xiamen, Fujian
  - 1st Aff Hosp of Shantou Univ /ID# 162968, Shantou, Guangdong
- Colombia (6):
  - Centro de Investigacion en Reumatologia y Especialidades Medicas- CIREEM SAS /ID# 143214, Bogota, Cundinamarca
  - Ctr Int de Reum del Caribe SAS /ID# 143211, Barranquilla
  - Riesgo de Fractura S.A - CAYRE /ID# 143212, Bogotá
  - Simedics IPS SAS /ID# 152572, Bogotá
  - Fund Inst de Reum F. Chalem /ID# 159544, Bogotá
  - Medicity S.A.S. /ID# 143213, Bucaramanga
- Croatia (4):
  - Klinicki bolnicki centar Split /ID# 143216, Split
  - Clinical Hospital Dubrava /ID# 143217, Zagreb
  - Medical Center Kuna-Peric /ID# 143218, Zagreb
  - Poliklinika Bonifarm /ID# 143215, Zagreb
- Czechia (11):
  - L.K.N. Arthrocentrum, s.r.o /ID# 143224, Hlučín, Moravskoslezský kraj
  - CTCenter MaVe, s.r.o. /ID# 143226, Olomouc, Olomoucký kraj
  - Nuselská poliklinika, Revmatologie /ID# 143232, Prague, Praha 4
  - Nuselská poliklinika, Revmatologie /ID# 143233, Prague, Praha 4
  - Thomayerova nemocnice /ID# 143228, Prague, Praha 4
  - PV MEDICAL Services s.r.o. /ID# 143234, Zlín, Zlín
  - Revmatologie, s.r.o. /ID# 143223, Brno
  - Revmatologie Bruntal, s.r.o /ID# 143220, Bruntál
  - RHEUMA s.r.o. /ID# 143230, Břeclav
  - Nemocnice Slany /ID# 143221, Slaný
  - Medical Plus, s.r.o. /ID# 143219, Uherské Hradište
- Estonia (4):
  - Center of Clinical and Basic Research /ID# 143239, Tallinn, Harju
  - Paernu Hospital /ID# 143238, Pärnu
  - East Tallinn Central Hospital /ID# 143240, Tallinn
  - North Estonian Medical Centre /ID# 145456, Tallinn
- Germany (6):
  - Uniklinik Koln /ID# 143248, Cologne, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet /ID# 145652, Herne, North Rhine-Westphalia
  - Praxis Walter, Rendsburg /ID# 143250, Rendsburg, Schleswig-Holstein
  - Rheumaforschungszentrum II /ID# 143247, Hamburg
  - Schoen Klinikum Hamburg Eilbek /ID# 143251, Hamburg
  - LMU Klinikum der Universität München /ID# 143249, Munich
- University General Hospital Attikon /ID# 143252, Athens, Attica, Greece
- Guatemala (5):
  - Clinicas Hospital Herrera Ller /ID# 153715, Guatemala City
  - Creer /Id# 153713, Guatemala City
  - Clin Especializada Med Interna /ID# 153716, Guatemala City
  - Clinica Medica Reumatologia /ID# 153714, Guatemala City
  - Clinica Medica Reumatologia /ID# 153931, Guatemala City
- Hong Kong (2):
  - Queen Mary Hospital /ID# 143255, Hong Kong
  - Tuen Mun Hospital /ID# 143256, Tuenmen
- Hungary (6):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 143258, Miskolc, Borsod-Abauj Zemplen county
  - Qualiclinic Kft. /ID# 143259, Budapest, Pest County
  - Markusovszky Egyetemi Oktatókórház /ID# 143261, Szombathely, Vas County
  - Hevizgyogyfurdo es Szent Andra /ID# 143257, Hévíz
  - Pest Megyei Flor Ferenc Korhaz /ID# 143260, Kistarcsa
  - Fejer Megyei Szent Gyorgy Korh /ID# 144724, Székesfehérvár
- St Vincent's University Hosp /ID# 143262, Dublin, Ireland
- Israel (3):
  - Barzilai Medical Center /ID# 144725, Ashkelon
  - Rambam Health Care Campus /ID# 143263, Haifa
  - Sheba Medical Center /ID# 145975, Ramat Gan
- Italy (4):
  - Istituto Clinico Humanitas /ID# 147531, Rozzano, Milano
  - Azienda Ospedaliera Luigi Sacc /ID# 143270, Milan
  - Fondazione IRCCS Policlinico /ID# 143265, Pavia
  - A.O.U.I. di Verona Policlinico /ID# 143266, Verona
- Japan (49):
  - Nagoya University Hospital /ID# 148031, Nagoya, Aichi-ken
  - NHO Toyohashi Medical Center /ID# 161033, Toyohashi, Aichi-ken
  - Teikyo University Chiba Medical Center /ID# 159618, Ichihara, Chiba
  - NHO Kyushu Medical Center /ID# 148263, Fukuoka, Fukuoka
  - NHO Kyushu Medical Center /ID# 148264, Fukuoka, Fukuoka
  - National Hospital Organization Asahikawa Medical Center /ID# 148021, Asahikawa, Hokkaido
  - Katayama Orthopedic Rheumatology Clinic /ID# 148029, Asahikawa, Hokkaido
  - Kobe University Hospital /ID# 153461, Kobe, Hyōgo
  - National Hospital Organization Sagamihara National Hospital /ID# 148019, Sagamihara-shi, Kanagawa
  - NHO Osaka Minami Med Ctr /ID# 148042, Osaka, Kawachinagano-shi
  - Bay Side Misato Medical Center /ID# 148256, Kochi, Kochi
  - Center for Arthritis and Clinical Rheumatology Matsubara Clinic /ID# 148254, Kumamoto, Kumamoto
  - Kumamoto Orthopaedic Hospital /ID# 148054, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital /ID# 148266, Kumamoto, Kumamoto
  - Sasebo Chuo Hospital /ID# 148261, Sasebo, Nagasaki
  - Nagaoka Red Cross Hospital /ID# 148018, Nagaoka-shi, Niigata
  - Japanese Red Cross Okayama Hospital /ID# 159619, Okayama, Okayama-ken
  - Kansai Medical University Hospital /ID# 159622, Hirakata-shi, Osaka
  - Osaka Medical College Hospital /ID# 159624, Takatsuki -shi, Osaka
  - Saitama Medical Center, Saitama Medical University /ID# 148015, Kawagoe-shi, Saitama
  - Jichi Medical University Hospital /ID# 159620, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital /ID# 148050, Bunkyo-ku, Tokyo
  - St.Luke's International Hospital /ID# 148041, Chuo-ku, Tokyo
  - Toho University Ohashi Medical Center /ID# 148027, Meguro-ku, Tokyo
  - Keio University Hospital /ID# 148057, Shinjuku-ku, Tokyo
  - Tokito Clinic Rheumatology and Orthopaedics Surgery /ID# 148052, Shimonoseki-shi, Yamaguchi
  - National Hospital Organization Beppu Medical Center /ID# 161058, Beppu
  - NHO Chiba-East-Hospital /ID# 148035, Chiba
  - Sugimoto Rheumatology and Internal Medicine Clinic /ID# 148047, Fukui
  - Shono Rheumatism Clinic /ID# 148046, Fukuoka
  - Matsubara Mayflower Hospital /ID# 148033, Katō
  - St. Mary's Hospital /ID# 148038, Kurume
  - Kagawa University Hospital /ID# 148016, Kyoto
  - Yu Family Clinic /ID# 148048, Miyagi
  - Daido Hospital /ID# 160868, Nagoya
  - Kondo Clinic for Ortho & Rheum /ID# 148032, Nagoya
  - Shirahama Hamayu Hospital /ID# 148253, Nishimura
  - Osaka City General Hospital /ID# 159617, Osaka
  - Oribe Clinic of Rheumatology and Internal Medicine /ID# 156035, Ōita
  - Sanuki Municipal Hospital /ID# 158842, Sanuki
  - Sagawa Akira Rheumatology Clin /ID# 148043, Sapporo
  - Sapporo City General Hospital /ID# 148037, Sapporo
  - Hokkaido University Hospital /ID# 148262, Sapporo
  - Hokkaido Medical Center for Rheumatic Diseases /ID# 148259, Sapporo
  - Azuma Rheumatology Clinic /ID# 161050, Sayama
  - Hikarigaoka Spellman Hospital /ID# 148020, Sendai
  - Takaoka Rheumatic Orthopedic Clinic /ID# 148022, Takaoka
  - National Hospital Organization Tokyo Medical Center /ID# 148040, Tokyo
  - National Hospital Organization Shimoshizu National Hospital /ID# 148258, Yotsukaidō
- Kazakhstan (4):
  - JSC Nat Scientific Med Res Ctr /ID# 143272, Astana
  - Karaganda State Medical Univ /ID# 153431, Karaganda
  - Semey State Medical University /ID# 152661, Semey
  - Regional Clinical Hospital /ID# 147173, Shymkent
- LTD M+M Centers /ID# 143279, Ādaži, Latvia
- Lithuania (3):
  - Hosp Lithuanian Univ Health Sc /ID# 143582, Kaunas, Kovno
  - Klaipeda University Hospital /ID# 143583, Klaipėda
  - Vilnius University Hospital /ID# 143584, Vilnius
- Mexico (7):
  - Clinstile, S.A. de C.V. /ID# 143591, Cuauhtémoc, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 153562, Mexico City, Mexico City
  - Invest y Biomed de Chihuahua /ID# 143595, Chihuahua City
  - RM Pharma Specialists, S.A de C.V /ID# 143593, Mexico City
  - Unidad de Investigacion de las Enfermedades Reumatologicas SA de CV /ID# 143592, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevención de Enfermedades Cardiova /ID# 143589, Mexico City
  - Centro Reumatologico de Queret /ID# 149493, Querétaro
- New Zealand (4):
  - Waikato Hospital /ID# 143602, Hamilton, Waikato Region
  - Middlemore Clinical Trials /ID# 143600, Auckland
  - Porter Rheumatology Ltd /ID# 143601, Nelson
  - Timaru Medical Specialists Ltd /ID# 143599, Timaru
- Poland (7):
  - Medyczne Centrum Hetmanska /ID# 144726, Poznan, Greater Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 143606, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne AMED /ID# 143604, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Warszawa /ID# 143608, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 143607, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp z o.o /ID# 143605, Katowice, Silesian Voivodeship
  - NZOZ Centrum Reumatologiczne /ID# 143603, Elblag, Warmian-Masurian Voivodeship
- Portugal (8):
  - Instituto Portugues De Reumatologia /ID# 148313, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 151009, Lisbon, Lisbon District
  - Centro Hospitalar De Vila Nova /ID# 143615, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 143613, Lisbon
  - Centro Hospitalar Baixo Vouga /ID# 153726, Porto
  - Centro Hospitalar de Sao Joao, EPE /ID# 153575, Porto
  - Unidade Local De Saude Do Alto Minho /ID# 143611, Viana do Castelo
  - Centro Hosp de Tondela-Viseu /ID# 143612, Viseu
- Puerto Rico (3):
  - Ponce School of Medicine /ID# 145657, Ponce
  - GCM Medical Group /ID# 143618, San Juan
  - School of Medicine University of Puerto Rico-Medical Sciences Campus /ID# 143619, San Juan
- Romania (6):
  - Spitalul Clinic Dr. I. Cantacuzino /ID# 143622, Bucharest, București
  - Spitalul Clinic Sf. Maria /ID# 143623, Bucharest
  - Spitalul Clinic Sf. Maria /ID# 143625, Bucharest
  - Spitalul Clinic Sf. Maria /ID# 143627, Bucharest
  - Spitalul Clinic de Recuperare /ID# 143620, Iași
  - Ecomed SRL /ID# 143629, Oradea
- Russia (14):
  - Family Outpatient clinic#4,LLC /ID# 151010, Korolev, Moscow
  - Clinical Hospital No.1 n.a. N.I.Pirogov /ID# 143641, Moscow, Moscow
  - LLC Medical Center /ID# 143647, Novosibirsk, Novosibirsk Oblast
  - LLC Novaya Klinika /ID# 143631, Pyatigorsk, Stavropol Kray
  - Kazan State Medical University /ID# 143645, Kazan', Tatarstan, Respublika
  - Tver Regional Clinical Hosp. /ID# 143639, Tver', Tver Oblast
  - Russian National Research Medi /ID# 143642, Moscow
  - Orenburg Regional Clinical Hos /ID# 143630, Orenburg
  - Republican Clin Hos n.a. Baran /ID# 143634, Petrozavodsk
  - Ryazan State Medical Universit /ID# 143646, Ryazan
  - Samara Regional Clinical Hosp /ID# 150928, Samara
  - Reg Clin Hosp n.a. Kuvatova G. /ID# 143632, Ufa
  - Ulyanovsk Regional Clin Hosp /ID# 143644, Ulyanovsk
  - Voronezh State Medical Univers /ID# 150926, Voronezh
- Serbia (3):
  - Clinical Center Serbia /ID# 143649, Belgrade, Beograd
  - Clinical Center Serbia /ID# 143650, Belgrade, Beograd
  - Special Hospital for Rheuma /ID# 143648, Novi Sad, Vojvodina
- Slovakia (11):
  - MEDMAN s.r.o. /ID# 143661, Martin
  - Reumatologická ambulancia Reum.hapi s.r.o. /ID# 143657, Nové Mesto nad Váhom
  - REUMACENTRUM s.r.o. /ID# 143653, Partizánske
  - Slovak research center Team Member, Thermium s.r.o. /ID# 143663, Pieštany
  - Slovak Research Center /ID# 143659, Púchov
  - TIMMED spol. s r.o. /ID# 143664, Stará Lubovna
  - Reumatologicka ambulancia, LER /ID# 143660, Topoľčany
  - MEDEOS s.r.o. /ID# 143656, Trenčín
  - REUMA-GLOBAL, s.r.o. /ID# 143655, Trnava
  - ALBAMED s.r.o. /ID# 143654, Zvolen
  - Reuma -MUDr. Maria Palasthyova /ID# 143662, Žiar nad Hronom
- Univ Medical Ctr Ljubljana /ID# 143667, Ljubljana, Slovenia
- South Africa (4):
  - Jakaranda Hosp, Emmed Research /ID# 143668, Pretoria, Gauteng
  - Jakaranda Hosp, Emmed Research /ID# 145976, Pretoria, Gauteng
  - Arthritis Clinical Research Tr /ID# 143670, Cape Town, Western Cape
  - Winelands Medical Research Ctr /ID# 143669, Stellenbosch, Western Cape
- Spain (6):
  - H. Un. Marques de Valdecilla /ID# 143671, Santander, Cantabria
  - Comple Hosp Univ de A Coruna /ID# 143672, A Coruña
  - Hospital Univ Vall d'Hebron /ID# 143675, Barcelona
  - Hospital Clin Univ San Carlos /ID# 143674, Madrid
  - Clinica Gaias /ID# 143673, Santiago de Compostela
  - Hosp Nuestra Senora Esperanza /ID# 143677, Santiago de Compostela
- HFR Fribourg - Hopital Canton /ID# 143700, Fribourg, Switzerland
- Taiwan (3):
  - China Medical University Hosp /ID# 143703, Taichung, Taichung
  - National Taiwan Univ Hosp /ID# 143702, Taipei City, Taipei
  - Dalin Tzu Chi General Hospital /ID# 153535, Dalin
- Tunisia (5):
  - Hopital Mongi Slim /ID# 152870, La Marsa
  - Institut Mohamed Kassab /ID# 152869, Manouba
  - Hopital Farhat Hached /ID# 152868, Sousse
  - Charles Nicolle Univ Hosp /ID# 152866, Tunis
  - Hospital La Rabta /ID# 152867, Tunis
- Turkey (Türkiye) (3):
  - Uludag Universitesi Ataturk Rehabilitasyon ve Uygulama Merkezi /ID# 143705, Osmangazi, Bursa
  - Izmir Tepecik Training and Research Hospital /ID# 157863, Konak, İzmir
  - Izmir Katip Celebi Ataturk Training & Research Hospital /ID# 143704, Izmir
- Ukraine (8):
  - Lviv Regional Clinical Hospita /ID# 154449, Lviv, Lviv Oblast
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 143714, Vinnytsia, Vinnytsia Oblast
  - Regional Clinical Hospital /ID# 152029, Ivano-Frankivsk
  - NSC-Strazhesko Ist Cardiology /ID# 152026, Kiev
  - LLC Revmocentr /ID# 143710, Kyiv
  - MNCE "Lviv City Clinical Hospital #4" /ID# 143711, Lviv
  - Odessa National Medical Univ /ID# 143715, Odesa
  - Zaporizhzhia Regional Clinical /ID# 143712, Zaporizhia
- United Kingdom (6):
  - Leicester Royal Infirmary /ID# 143718, Leicester, England
  - Whipps Cross Univ Hospital /ID# 143721, London, London, City of
  - Western General Hospital /ID# 144431, Edinburgh
  - Chapel Allerton Hospital /ID# 143717, Leeds
  - Queen Alexandra Hospital /ID# 143722, Portsmouth
  - Southampton General Hospital /ID# 143716, Southampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] van Vollenhoven R, Takeuchi T, Pangan AL, Friedman A, Mohamed MF, Chen S, Rischmueller M, Blanco R, Xavier RM, Strand V. Efficacy and Safety of Upadacitinib Monotherapy in Methotrexate-Naive Patients With Moderately-to-Severely Active Rheumatoid Arthritis (SELECT-EARLY): A Multicenter, Multi-Country, Randomized, Double-Blind, Active Comparator-Controlled Trial. Arthritis Rheumatol. 2020 Oct;72(10):1607-1620. doi: 10.1002/art.41384. Epub 2020 Sep 8. PMID 32638504
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] van Vollenhoven R, Strand V, Takeuchi T, Chavez N, Walter PM, Singhal A, Swierkot J, Khan N, Bu X, Li Y, Penn SK, Camp HS, Aelion J. Upadacitinib monotherapy versus methotrexate monotherapy in patients with rheumatoid arthritis: efficacy and safety through 5 years in the SELECT-EARLY randomized controlled trial. Arthritis Res Ther. 2024 Jul 29;26(1):143. doi: 10.1186/s13075-024-03358-x. PMID 39075620
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Buch MH, Tanaka Y, Citera G, Bahlas S, Wong E, Song Y, Zueger P, Ali M, Strand V. Routine Assessment of Patient Index Data 3 (RAPID3) in Patients with Rheumatoid Arthritis Treated with Long-Term Upadacitinib Therapy in Five Randomized Controlled Trials. Rheumatol Ther. 2022 Dec;9(6):1517-1529. doi: 10.1007/s40744-022-00483-4. Epub 2022 Sep 20. PMID 36125701
- [Derived] Peterfy CG, Strand V, Friedman A, Hall S, Mysler E, Durez P, Baraliakos X, Enejosa JV, Shaw T, Li Y, Chen S, Song IH. Inhibition of structural joint damage progression with upadacitinib in rheumatoid arthritis: 1-year outcomes from the SELECT phase 3 program. Rheumatology (Oxford). 2022 Aug 3;61(8):3246-3256. doi: 10.1093/rheumatology/keab861. PMID 34897366
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Strand V, Tundia N, Wells A, Buch MH, Radominski SC, Camp HS, Friedman A, Suboticki JL, Dunlap K, Goldschmidt D, Bergman M. Upadacitinib monotherapy improves patient-reported outcomes in rheumatoid arthritis: results from SELECT-EARLY and SELECT-MONOTHERAPY. Rheumatology (Oxford). 2021 Jul 1;60(7):3209-3221. doi: 10.1093/rheumatology/keaa770. PMID 33313898
- [Derived] Cohen SB, van Vollenhoven RF, Winthrop KL, Zerbini CAF, Tanaka Y, Bessette L, Zhang Y, Khan N, Hendrickson B, Enejosa JV, Burmester GR. Safety profile of upadacitinib in rheumatoid arthritis: integrated analysis from the SELECT phase III clinical programme. Ann Rheum Dis. 2021 Mar;80(3):304-311. doi: 10.1136/annrheumdis-2020-218510. Epub 2020 Oct 28. PMID 33115760
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 236 sites in 43 countries. The study included 2 periods and a Japan sub-study. The global study analysis included participants from Japan, but excluded the upadacitinib 7.5 mg group. The Japan sub-study included all participants from Japan, including the upadacitinib 7.5 mg group.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to Groups 1, 3, and 4 below, except for participants in Japan who were randomized in a 1:2:1:1 ratio to Groups 1, 2, 3, and 4. Randomization was stratified by geographic region.
  Efficacy analyses were conducted separately for the Japan sub-study.
Groups:
- Methotrexate: Group 1 participants received up to 20 mg methotrexate orally per week (15 mg/week in China and Japan) and placebo to upadacitinib once a day (QD) for 48 weeks during Period 1.
  Participants who did not achieve Clinical Remission (CR) based on clinical disease activity index (CDAI) score (CDAI ≤ 2.8) and did not achieve a ≥ 20% improvement from Baseline in both tender joint count (TJC) and swollen joint count (SJC) at Week 26 were re-randomized in a 1:1 ratio to receive rescue therapy with upadacitinib 15 mg or 30 mg QD (or in a 1:1:1 ratio to receive upadacitinib 7.5 mg, 15 mg, or 30 mg QD for participants in Japan) in addition to methotrexate.
  In Period 2 (Weeks 48 to 260) participants continued to receive the treatment they were assigned at the end of Period 1.
- Upadacitinib 7.5 mg: Group 2 participants (Japan only) received 7.5 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
  Participants who did not achieve CR based on CDAI and did not achieve a ≥ 20% improvement from Baseline in both TJC and SJC at Week 26 received rescue treatment with methotrexate 7.5 mg/week in addition to continuing to receive upadacitinib 7.5 mg QD.
  In Period 2 participants continued to receive the treatment they were assigned at the end of Period 1.
- Upadacitinib 15 mg: Group 3 participants received 15 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
  Participants who did not achieve CR based on CDAI and did not achieve a ≥ 20% improvement from Baseline in both TJC and SJC at Week 26 received rescue treatment with methotrexate 10 mg/week (7.5 mg for China and Japan) in addition to continuing to receive upadacitinib 15 mg QD.
  In Period 2 participants continued to receive the treatment they were assigned at the end of Period 1 up to Week 260.
- Upadacitinib 30 mg: Group 4 participants received 30 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
  Participants who did not achieve CR by CDAI and did not achieve a ≥ 20% improvement from Baseline in both TJC and SJC at Week 26 received rescue treatment with methotrexate 10 mg/week (7.5 mg for China and Japan) in addition to continuing to receive upadacitinib 30 mg QD.
  In Period 2 participants continued to receive the treatment they were assigned at the end of Period 1. Starting with Protocol Amendment 6 participants were switched to receive open-label upadacitinib 15 mg QD.
Period: Period 1 (Weeks 1 to 48)
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 315 | 55 | 317 | 315
Received Study Drug | 314 | 55 | 317 | 314
Global Analysis Population (Participants enrolled in the methotrexate, upadacitinib 15 mg and 30 mg treatment groups) | 314 (Includes 28 participants in the Japan sub-study) | 0 | 317 (Includes 27 participants in the Japan sub-study) | 314 (Includes 28 participants in the Japan sub-study)
Japan Sub-study (Participants in the methotrexate, upadacitinib 7.5, 15, and 30 mg treatment groups enrolled in Japan) | 28 | 55 | 27 | 28
Completed Week 24 Study Drug | 268 | 51 | 290 | 282
Received Combination Rescue Therapy at Week 26 | 37 (Combination therapy includes the addition of upadacitinib to methotrexate. Participants with inadequate response were randomized equally to receive upadacitinib 7.5 mg (Japan only), 15 mg or 30 mg QD in addition to methotrexate. One participant received upadacitinib 7.5 mg; 18 participants received upadacitinib 15 mg; 18 participants received upadacitinib 30 mg.) | 3 (Combination therapy includes the addition of methotrexate to upadacitinib 7.5 mg.) | 19 (Combination therapy includes the addition of methotrexate to upadacitinib 15 mg.) | 9 (Combination therapy includes the addition of methotrexate to upadacitinib 30 mg.)
Completed (Completed Week 48) | 256 | 51 | 277 | 271
Not Completed | 59 | 4 | 40 | 44
Not completed — Adverse Event | 15 | 3 | 18 | 11
Not completed — Withdrawal by Subject | 22 | 0 | 12 | 20
Not completed — Lost to Follow-up | 4 | 0 | 6 | 5
Not completed — Lack of Efficacy | 12 | 0 | 2 | 4
Not completed — Other | 5 | 1 | 2 | 3
Not completed — Not Dosed | 1 | 0 | 0 | 1
Period: Period 2 (Weeks 48 to 260)
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started (Nine participants who completed Period 1 opted not to enter Period 2.) | 253 | 50 | 275 | 268
Received Study Drug | 242 | 48 | 273 | 260
Completed | 163 | 40 | 217 | 187
Not Completed | 90 | 10 | 58 | 81
Not completed — Adverse Event | 16 | 4 | 11 | 26
Not completed — Withdrawal by Subject | 32 | 5 | 23 | 27
Not completed — Lost to Follow-up | 17 | 0 | 10 | 6
Not completed — Lack of Efficacy | 11 | 0 | 1 | 1
Not completed — Coronavirus Disease of 2019 (COVID-19) Infection | 0 | 0 | 0 | 3
Not completed — COVID-19 Logistic Restrictions | 0 | 0 | 2 | 1
Not completed — Other | 14 | 1 | 11 | 17

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Methotrexate: Participants received up to 20 mg methotrexate orally per week and placebo to upadacitinib once a day for 48 weeks during Period 1.
- Upadacitinib 7.5 mg: Participants received 7.5 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
- Upadacitinib 15 mg: Participants received 15 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
- Upadacitinib 30 mg: Participants received 30 mg upadacitinib orally once a day and placebo to methotrexate once a week for 48 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 314 | 55 | 317 | 314 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.89) | 59.7 (13.8) | 51.9 (12.58) | 54.9 (12.58) | 53.7 (12.86)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 50 | 5 | 60 | 34 | 149
  40 - 65 years | 206 | 25 | 204 | 212 | 647
  ≥ 65 years | 58 | 25 | 53 | 68 | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 36 | 241 | 240 | 757
  Male | 74 | 19 | 76 | 74 | 243
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 0 | 107 | 107 | 316
  Not Hispanic or Latino | 212 | 55 | 210 | 207 | 684
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 256 | 0 | 256 | 254 | 766
  Black or African American | 12 | 0 | 8 | 13 | 33
  American Indian/Alaska Native | 2 | 0 | 8 | 7 | 17
  Native Hawaiian or other Pacific Islander | 2 | 0 | 3 | 1 | 6
  Asian | 37 | 55 | 35 | 34 | 161
  Multiple | 5 | 0 | 7 | 5 | 17
Geographic Region [Count of Participants; unit: Participants]
  North America | 46 | 0 | 48 | 46 | 140
  South/Central America | 90 | 0 | 91 | 91 | 272
  Western Europe | 37 | 0 | 36 | 36 | 109
  Eastern Europe | 85 | 0 | 87 | 87 | 259
  Asia-Japan | 28 | 55 | 27 | 28 | 138
  Asia - China | 1 | 0 | 1 | 1 | 3
  Asia - Other | 3 | 0 | 4 | 2 | 9
  Other | 24 | 0 | 23 | 23 | 70
Duration of Rheumatoid Arthritis Diagnosis [Mean (Standard Deviation); unit: years] | 2.6 (5.14) | 2.3 (5.77) | 2.9 (5.38) | 2.8 (5.63) | 2.7 (5.40)
Tender Joint Count [Mean (Standard Deviation); unit: tender joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  tender joints | 26.4 (16.15) | 18.0 (11.75) | 25.4 (14.42) | 25.2 (14.99) | 25.3 (15.12)
Swollen Joint Count [Mean (Standard Deviation); unit: swollen joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  swollen joints | 16.9 (10.58) | 14.7 (8.24) | 16.9 (10.35) | 15.7 (9.71) | 16.4 (10.13)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain." Population: Participants with available data
  mm
    number analyzed (Participants) | 314 | 55 | 317 | 311 | 997
    (all) | 65.7 (21.46) | 64.1 (21.20) | 68.4 (20.60) | 65.3 (21.51) | 66.3 (21.21)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 314 | 55 | 317 | 311 | 997
    (all) | 65.8 (21.45) | 64.1 (21.36) | 66.6 (22.01) | 64.9 (21.63) | 65.7 (21.66)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 299 | 54 | 301 | 304 | 958
    (all) | 68.7 (16.45) | 63.3 (19.34) | 67.1 (17.00) | 65.3 (16.60) | 66.8 (16.89)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 314 | 55 | 317 | 311 | 997
    (all) | 1.6 (0.67) | 1.3 (0.62) | 1.6 (0.67) | 1.5 (0.66) | 1.6 (0.66)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 21.2 (22.05) | 18.5 (17.55) | 23.0 (27.37) | 19.4 (22.59) | 21.0 (23.84)
Disease Activity Score 28 Based on CRP (DAS28[CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 314 | 55 | 317 | 311 | 997
    (all) | 5.9 (0.97) | 5.5 (0.90) | 5.9 (0.97) | 5.8 (1.02) | 5.8 (0.99)
Modified Total Sharp Score (mTSS) [Mean (Standard Deviation); unit: units on a scale] — The mTSS measures the level of joint damage from radiographs of the hands and feet, calculated as the sum of the total joint erosion score and total joint space narrowing (JSN) score and ranges from 0 (normal) to 448 (worst). Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 309 | 55 | 309 | 309 | 982
    (all) | 13.3 (30.55) | 15.9 (39.10) | 18.1 (38.15) | 17.2 (38.25) | 16.1 (36.02)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12 - Global Analysis
Description: The primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was ACR 50% response (ACR50) at Week 12. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
  The global analysis includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 28.3 [23.4 to 33.3] | 52.1 [46.6 to 57.5] | 56.4 [50.9 to 61.9]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; For the global analysis, comparisons of the primary and key secondary efficacy endpoints were made between the upadacitinib 15 mg and 30 mg groups versus the methotrexate group; Test type: Superiority — The overall type I error rate of the primary and ranked key secondary endpoints for the two upadacitinib doses (15 mg and 30 mg) was controlled using a graphical multiple testing procedure defined separately for US/FDA, European Union/European Medicines Agency and Japan/Pharmaceuticals and Medical Devices Agency regulatory purposes; p < 0.001, Cochran-Mantel-Haenszel — The adjusted p-value under multiplicity control is reported, with significance achieved if the adjusted p-value is less than 0.05; Cochran-Mantel-Haenszel test adjusting for geographic region (North America, South/central America, Western Europe, Eastern Europe, Asia/other); Response Rate Difference = 23.7, 95% CI 2-sided [16.3 to 31.1] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 28.0, 95% CI 2-sided [20.6 to 35.4] — Response Rate Difference = Upadacitinib - Methotrexate

2. Primary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 24 - Global Analysis
Description: The primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was clinical remission, based on a Disease Activity Score 28 (DAS28)-CRP score of < 2.6 at Week 24.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Week 24
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 24 or for whom DAS28 data were missing at Week 24 were considered non-responders.
  The global analysis includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 18.5 [14.2 to 22.8] | 48.3 [42.8 to 53.8] | 50.0 [44.5 to 55.5]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 29.8, 95% CI 2-sided [22.8 to 36.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 31.5, 95% CI 2-sided [24.5 to 38.5] — Response Rate Difference = Upadacitinib - Methotrexate

3. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12 - Global Analysis
Description: The primary endpoint for Japan/Pharmaceuticals and Medical Devices Agency (PMDA) regulatory purposes was ACR 20% response (ACR20) at Week 12. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 54.1 [48.6 to 59.7] | 75.7 [71.0 to 80.4] | 77.1 [72.4 to 81.7]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 21.6, 95% CI 2-sided [14.3 to 28.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 22.9, 95% CI 2-sided [15.7 to 30.1] — Response Rate Difference = Upadacitinib - Methotrexate

4. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 24 - Global Analysis
Description: The second primary endpoint for Japan/PMDA regulatory purposes was change from baseline in mTSS at Week 24.
  The mTSS measures the level of joint damage from radiographs of the hands and feet. Joint erosion and joint space narrowing (JSN) were assessed by two independent, blinded readers.
  Joint erosion was assessed in 16 joints in each hand/wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 280 (worst).
  JSN was assessed in 15 joints of each hand and wrist, and 6 joints of each foot, including subluxation, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 168 (worst).
  The mTSS is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 448 (worst). A change from Baseline greater than 0 indicates progression.
Time Frame: Baseline to Week 24
Population: Full analysis set participants with available data at Baseline; linear extrapolation was used for participants who discontinued prior to Week 24 or for whom x-ray data were missing at Week 24.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 264 | 279 | 270
units on a scale | 0.67 [0.43 to 0.90] | 0.14 [-0.09 to 0.37] | 0.07 [-0.16 to 0.31]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of covariance (ANCOVA) model with treatment, geographic region as fixed factors and baseline value as the covariate; Least Squares (LS) Mean Difference = -0.53, 95% CI 2-sided [-0.85 to -0.20] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.59, 95% CI 2-sided [-0.91 to -0.27] — Difference = Upadacitinib - Methotrexate

5. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Week 12 - Global Analysis
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline to Week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing post-baseline data.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 312 | 317 | 310
scores on a scale | -1.85 [-2.00 to -1.69] | -2.73 [-2.87 to -2.58] | -2.85 [-3.00 to -2.70]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of the primary and ranked key secondary endpoints for the two doses was controlled using a graphical multiple testing procedure. This endpoint was a ranked key secondary endpoint for US/FDA and Japan/PMDA regulatory purposes; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.88, 95% CI 2-sided [-1.09 to -0.67]
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -1.01, 95% CI 2-sided [-1.21 to -0.80] — Difference = Upadacitinib - Methotrexate

6. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 - Global Analysis
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline to week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing data.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 313 | 317 | 310
scores on a scale | -0.49 [-0.55 to -0.42] | -0.83 [-0.90 to -0.76] | -0.86 [-0.93 to -0.79]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.34, 95% CI 2-sided [-0.44 to -0.25] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.37, 95% CI 2-sided [-0.47 to -0.28] — Difference = Upadacitinib - Methotrexate

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12 - Global Analysis
Description: The DAS28(CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28(CRP) score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 28.3 [23.4 to 33.3] | 53.3 [47.8 to 58.8] | 54.8 [49.3 to 60.3]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 25.0, 95% CI 2-sided [17.6 to 32.4] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Chi-squared, Corrected — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 26.4, 95% CI 2-sided [19.0 to 33.9]; Response Rate Difference = Upadacitinib - Methotrexate

8. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12 - Global Analysis
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline to week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 311 | 315 | 311
scores on a scale | 5.74 [4.84 to 6.64] | 9.99 [9.11 to 10.88] | 10.08 [9.19 to 10.98]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = 4.25, 95% CI 2-sided [3.00 to 5.50] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = 4.34, 95% CI 2-sided [3.09 to 5.59] — Difference = Upadacitinib - Methotrexate

9. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Week 24 - Global Analysis
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 312 | 317 | 310
scores on a scale | -2.15 [-2.31 to -1.99] | -3.07 [-3.21 to -2.92] | -3.34 [-3.49 to -3.19]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of the primary and ranked key secondary endpoints for the two doses was controlled using a graphical multiple testing procedure. This endpoint was a ranked key secondary endpoint for EU/EMA regulatory purposes; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.92, 95% CI 2-sided [-1.12 to -0.71] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -1.19, 95% CI 2-sided [-1.40 to -0.99] — Difference = Upadacitinib - Methotrexate

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 24 - Global Analysis
Description: as for outcome 6
Time Frame: Baseline to Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 313 | 317 | 310
scores on a scale | -0.60 [-0.67 to -0.52] | -0.87 [-0.94 to -0.80] | -0.91 [-0.98 to -0.84]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.27, 95% CI 2-sided [-0.37 to -0.17] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = -0.31, 95% CI 2-sided [-0.41 to -0.21] — Difference = Upadacitinib - Methotrexate

11. Secondary Outcome: Percentage of Participants With an ACR50 Response at Week 24 - Global Analysis
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 24 or for whom ACR data were missing at Week 24 were considered non-responders.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 33.4 [28.2 to 38.7] | 60.3 [54.9 to 65.6] | 65.6 [60.4 to 70.9]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 26.8, 95% CI 2-sided [19.3 to 34.3] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 32.2, 95% CI 2-sided [24.8 to 39.6] — Response Rate Difference = Upadacitinib - Methotrexate

12. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 24 - Global Analysis
Description: as for outcome 7
Time Frame: Week 24
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 24 or for whom DAS28 data were missing at Week 24 were considered non-responders.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 32.2 [27.0 to 37.3] | 59.9 [54.5 to 65.3] | 65.0 [59.7 to 70.2]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 27.8, 95% CI 2-sided [20.3 to 35.2] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 32.8, 95% CI 2-sided [25.4 to 40.2] — Response Rate Difference = Upadacitinib - Methotrexate

13. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 24 - Global Analysis
Description: as for outcome 8
Time Frame: Baseline to Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 313 | 315 | 312
scores on a scale | 6.97 [6.03 to 7.91] | 10.70 [9.76 to 11.63] | 11.39 [10.42 to 12.36]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = 3.72, 95% CI 2-sided [2.42 to 5.03] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, ANCOVA — The nominal p-value is reported; ANCOVA model with treatment and geographic region as fixed factors and Baseline value as the covariate; LS Mean Difference = 4.42, 95% CI 2-sided [3.12 to 5.72] — Difference = Upadacitinib - Methotrexate

14. Secondary Outcome: Percentage of Participants With No Radiographic Progression at Week 24 - Global Analysis
Description: No radiographic progression is defined as a change from Baseline in mTSS ≤ 0. The mTSS measures the level of joint damage from radiographs of the hands and feet. Joint erosion and joint space narrowing (JSN) were assessed by two independent, blinded readers.
  Joint erosion severity was assessed in 16 joints in each hand and wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 280 (worst).
  Joint space narrowing (JSN) was assessed in 15 joints of each hand and wrist, and 6 joints of each foot, including subluxation, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 168 (worst).
  The mTSS is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 448 (worst).
Time Frame: Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 264 | 279 | 270
percentage of participants | 77.7 [72.6 to 82.7] | 87.5 [83.6 to 91.3] | 89.3 [85.6 to 93.0]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.002, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 9.8, 95% CI 2-sided [3.5 to 16.2] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 11.6, 95% CI 2-sided [5.4 to 17.8] — Response Rate Difference = Upadacitinib - Methotrexate

15. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12 - Global Analysis
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
  The global analysis population includes participants enrolled under the methotrexate and upadacitinib 15 mg and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 14.0 [10.2 to 17.9] | 32.5 [27.3 to 37.6] | 36.9 [31.6 to 42.3]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 18.5, 95% CI 2-sided [12.1 to 24.9] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 22.9, 95% CI 2-sided [16.4 to 29.5] — Response Rate Difference = Upadacitinib - Methotrexate

16. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 24 - Global Analysis
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 58.6 [53.2 to 64.0] | 78.9 [74.4 to 83.4] | 78.0 [73.4 to 82.6]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 20.3, 95% CI 2-sided [13.2 to 27.3] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 19.4, 95% CI 2-sided [12.3 to 26.5] — Response Rate Difference = Upadacitinib - Methotrexate

17. Secondary Outcome: Percentage of Participants With an ACR70 Response at Week 24 - Global Analysis
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 314 | 317 | 314
percentage of participants | 18.5 [14.2 to 22.8] | 44.5 [39.0 to 49.9] | 49.7 [44.2 to 55.2]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 26.0, 95% CI 2-sided [19.1 to 33.0] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The nominal p-value is reported; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 31.2, 95% CI 2-sided [24.2 to 38.2] — Response Rate Difference = Upadacitinib - Methotrexate

18. Secondary Outcome: Percentage of Participants With an ACR20 Response at Week 12 - Japan Sub-study
Description: as for outcome 16
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
  The Japan sub-study analysis includes participants enrolled in Japan under the methotrexate and upadacitinib 7.5 mg, 15 mg, and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
percentage of participants | 57.1 [38.8 to 75.5] | 85.5 [76.1 to 94.8] | 85.2 [71.8 to 98.6] | 78.6 [63.4 to 93.8]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority — For the Japan sub-study, no multiplicity adjustments were applied and only nominal p-values were provided for all efficacy analyses; p = 0.004, Chi-squared; Response Rate Difference = 28.3, 95% CI 2-sided [7.7 to 48.9] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p = 0.022, Chi-squared; Response Rate Difference = 28.0, 95% CI 2-sided [5.3 to 50.7] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p = 0.086, Chi-squared; Response Rate Difference = 21.4, 95% CI 2-sided [-2.4 to 45.2] — Response Rate Difference = Upadacitinib - Methotrexate

19. Secondary Outcome: Percentage of Participants With an ACR50 Response at Week 12 - Japan Sub-study
Description: as for outcome 11
Time Frame: Baseline and Week 12
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
percentage of participants | 21.4 [6.2 to 36.6] | 60.0 [47.1 to 72.9] | 66.7 [48.9 to 84.4] | 71.4 [54.7 to 88.2]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 38.6, 95% CI 2-sided [18.6 to 58.5] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 45.2, 95% CI 2-sided [21.8 to 68.6] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 50.0, 95% CI 2-sided [27.4 to 72.6] — Response Rate Difference = Upadacitinib - Methotrexate

20. Secondary Outcome: Percentage of Participants With an ACR70 Response at Week 12 - Japan Sub-study
Description: as for outcome 15
Time Frame: Baseline and Week 12
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
percentage of participants | 0.0 [0.0 to 0.0] | 34.5 [22.0 to 47.1] | 51.9 [33.0 to 70.7] | 64.3 [46.5 to 82.0]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 34.5, 95% CI 2-sided [22.0 to 47.1] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 51.9, 95% CI 2-sided [33.0 to 70.7] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 64.3, 95% CI 2-sided [46.5 to 82.0] — Response Rate Difference = Upadacitinib - Methotrexate

21. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Week 12 - Japan Sub-study
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing post-baseline data.
  The Japan sub-study analysis includes participants enrolled in Japan under the methotrexate and upadacitinib 7.5 mg, 15 mg, and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
scores on a scale | -1.42 [-1.82 to -1.03] | -2.86 [-3.14 to -2.58] | -3.28 [-3.68 to -2.89] | -3.34 [-3.74 to -2.95]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -1.43, 95% CI 2-sided [-1.92 to -0.95] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -1.86, 95% CI 2-sided [-2.42 to -1.30] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -1.92, 95% CI 2-sided [-2.48 to -1.36] — Difference = Upadacitinib - Methotrexate

22. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 - Japan Sub-study
Description: as for outcome 6
Time Frame: Baseline to week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing data.
  The Japan sub-study analysis includes participants enrolled in Japan under the methotrexate and upadacitinib 7.5 mg, 15 mg, and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
scores on a scale | -0.20 [-0.37 to -0.04] | -0.75 [-0.86 to -0.63] | -0.95 [-1.12 to -0.78] | -0.95 [-1.12 to -0.79]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -0.54, 95% CI 2-sided [-0.75 to -0.34] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -0.75, 95% CI 2-sided [-0.99 to -0.51] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -0.75, 95% CI 2-sided [-0.99 to -0.51] — Difference = Upadacitinib - Methotrexate

23. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12 - Japan Sub-study
Description: as for outcome 8
Time Frame: Baseline to Week 12
Population: as for outcome 22
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
scores on a scale | 2.87 [0.56 to 5.18] | 8.84 [7.18 to 10.50] | 10.79 [8.48 to 13.09] | 9.63 [7.13 to 12.13]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = 5.97, 95% CI 2-sided [3.15 to 8.80] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = 7.92, 95% CI 2-sided [4.66 to 11.19] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = 6.76, 95% CI 2-sided [3.33 to 10.20] — Difference = Upadacitinib - Methotrexate

24. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12 - Japan Sub-study
Description: as for outcome 7
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
  The Japan sub-study analysis includes participants enrolled in Japan under the methotrexate and upadacitinib 7.5 mg, 15 mg, and 30 mg treatment groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
percentage of participants | 17.9 [3.7 to 32.0] | 69.1 [56.9 to 81.3] | 77.8 [62.1 to 93.5] | 78.6 [63.4 to 93.8]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 51.2, 95% CI 2-sided [32.5 to 70.0] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 59.9, 95% CI 2-sided [38.8 to 81.1] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 60.7, 95% CI 2-sided [39.9 to 81.5] — Response Rate Difference = Upadacitinib - Methotrexate

25. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 24 - Japan Sub-study
Description: The DAS28(CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Week 24
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 28 | 55 | 27 | 28
percentage of participants | 17.9 [3.7 to 32.0] | 67.3 [54.9 to 79.7] | 70.4 [53.1 to 87.6] | 82.1 [68.0 to 96.3]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 49.4, 95% CI 2-sided [30.6 to 68.3] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 52.5, 95% CI 2-sided [30.2 to 74.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Chi-squared; Response Rate Difference = 64.3, 95% CI 2-sided [44.2 to 84.3] — Response Rate Difference = Upadacitinib - Methotrexate

26. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 24 - Japan Sub-study
Description: The mTSS measures the level of joint damage from radiographs of the hands and feet. Joint erosion and joint space narrowing (JSN) were assessed by two independent, blinded readers.
  Joint erosion was assessed in 16 joints in each hand/wrist and 6 joints in each foot. Each joint was scored from 0 (no erosion) to 5 for hands/wrists or to 10 for feet (complete collapse). The total erosion score ranges from 0 to 280 (worst).
  JSN was assessed in 15 joints of each hand and wrist, and 6 joints of each foot, including subluxation, from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation). The total JSN score ranges from 0 to 168 (worst).
  The mTSS is the sum of the joint erosion and JSN scores and ranges from 0 (normal) to 448 (worst). A change from Baseline greater than 0 indicates progression.
Time Frame: Baseline to Week 24
Population: Full analysis set participants with available data at Baseline; linear extrapolation was used for participants who discontinued prior to Week 24 or for whom x-ray data were missing at Week 24.
  The Japan sub-study analysis includes participants enrolled in Japan under the methotrexate and upadacitinib 7.5 mg, 15 mg, and 30 mg treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 26 | 51 | 26 | 24
units on a scale | 2.64 [1.19 to 4.09] | 0.95 [-0.09 to 1.98] | 0.24 [-1.21 to 1.69] | 0.19 [-1.31 to 1.70]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.063, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -1.69, 95% CI 2-sided [-3.47 to 0.09] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p = 0.022, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -2.40, 95% CI 2-sided [-4.45 to -0.35] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p = 0.022, ANOVA; ANOVA model with Baseline value as covariate; LS Mean Difference = -2.45, 95% CI 2-sided [-4.54 to -0.35] — Difference = Upadacitinib - Methotrexate

27. Secondary Outcome: Percentage of Participants With No Radiographic Progression at Week 24 - Japan Sub-study
Description: as for outcome 14
Time Frame: Week 24
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 26 | 51 | 26 | 24
percentage of participants | 46.2 [27.0 to 65.3] | 82.4 [71.9 to 92.8] | 80.8 [65.6 to 95.9] | 79.2 [62.9 to 95.4]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.001, Chi-squared; Response Rate Difference = 36.2, 95% CI 2-sided [14.4 to 58.0] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p = 0.010, Chi-squared; Response Rate Difference = 34.6, 95% CI 2-sided [10.2 to 59.0] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 3: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p = 0.016, Chi-squared; Response Rate Difference = 33.0, 95% CI 2-sided [7.9 to 58.1] — Response Rate Difference = Upadacitinib - Methotrexate

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose, maximum of 264 weeks; Adverse events (AEs) are reported for Weeks 1 to 24, Weeks 1 to 260, and After Switch for participants who transitioned from upadacitinib 30 mg QD to 15 mg QD after implementation of Protocol Amendment 6 in December 2019.
Description: In Weeks 1 to 24 all participants received monotherapy. For Weeks 1 to 260 and After Switch, AEs are reported for the following:
  * Monotherapy: includes participants receiving monotherapy until the end of study or until rescue treatment was initiated.
  * All upadacitinib: includes any exposure to upadacitinib, alone or in addition to methotrexate or csDMARD after rescue, including participants originally assigned to methotrexate who were rescued with methotrexate + upadacitinib at Week 26.
Groups:
- Weeks 1-24: Methotrexate Monotherapy: Participants received up to 20 mg methotrexate orally per week (15 mg/week in China and Japan) and placebo to upadacitinib QD for 24 weeks during Period 1.
- Weeks 1-24: Upadacitinib 7.5 mg Monotherapy: Participants received 7.5 mg upadacitinib orally once a day and placebo to methotrexate once a week for 24 weeks in Period 1.
- Weeks 1-24: Upadacitinib 15 mg Monotherapy: Participants received 15 mg upadacitinib orally once a day and placebo to methotrexate once a week for 24 weeks in Period 1.
- Weeks 1-24: Upadacitinib 30 mg Monotherapy: Participants received 30 mg upadacitinib orally once a day and placebo to methotrexate once a week for 24 weeks in Period 1.
- Weeks 1-260: Methotrexate Monotherapy: Participants received up to 20 mg methotrexate orally per week (15 mg/week in China and Japan) for 260 weeks. Includes events up until the addition of upadacitinib for participants who were rescued at Week 26.
- Weeks 1-260: Upadacitinib 7.5 mg Monotherapy: Participants received 7.5 mg upadacitinib monotherapy once a day for 260 weeks. Includes events up until the addition of methotrexate or addition of background conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) for participants who received rescue.
- Weeks 1-260: Upadacitinib 15 mg Monotherapy: Participants received 15 mg upadacitinib monotherapy once a day for 260 weeks. Includes events up until the addition of methotrexate or addition of background csDMARD for participants who received rescue.
- Weeks 1-260/Switch: Upadacitinib 30 mg Monotherapy: Participants received 30 mg upadacitinib monotherapy once a day for 260 weeks or until implementation of Protocol Amendment 6 (December 2019) when they were switched to upadacitinib 15 mg. Includes events up until the addition of methotrexate or addition of background csDMARD for participants who received rescue, or up until the switch to upadacitinib 15 mg.
- Weeks 1-260: Any Upadacitinib 7.5 mg: Participants originally randomized to upadacitinib 7.5 mg received upadacitinib 7.5 mg QD for up to 260 weeks, including events after the addition of rescue therapy. Participants originally randomized to methotrexate and rescued at Week 26 to methotrexate plus upadacitinib 7.5 mg received upadacitinib 7.5 mg QD from Week 26 to Week 260.
- Weeks 1-260: Any Upadacitinib 15 mg: Participants originally randomized to upadacitinib 15 mg received upadacitinib 15 mg QD for up to 260 weeks, including events after the addition of rescue therapy. Participants originally randomized to methotrexate and rescued at Week 26 to methotrexate plus upadacitinib 15 mg received upadacitinib 15 mg QD from Week 26 to Week 260.
- Weeks 1-260/Switch: Any Upadacitinib 30 mg: Participants originally randomized to upadacitinib 30 mg received upadacitinib 30 mg QD for up to 260 weeks or until implementation of Protocol Amendment 6 (December 2019) when they were switched to upadacitinib 15 mg, including events after the addition of rescue therapy. Participants originally randomized to methotrexate and rescued at Week 26 to methotrexate plus upadacitinib 30 mg received upadacitinib 30 mg QD from Week 26 to Week 260 or until implementation of Protocol Amendment 6 when they were switched to methotrexate plus upadacitinib 15 mg. Includes events up until the switch to upadacitinib 15 mg.
- After Switch: Upadacitinib 15 mg Monotherapy: Participants who were receiving upadacitinib 30 mg QD monotherapy in Period 2 were switched to receive upadacitinib 15 mg QD monotherapy after implementation of Protocol Amendment 6 (December 2019) up to Week 260.
- After Switch: Any Upadacitinib 15 mg: Participants who were receiving any upadacitinib 30 mg QD (monotherapy or in combination with methotrexate or csDMARD after rescue) in Period 2 were switched to receive upadacitinib 15 mg QD (monotherapy or in combination with methotrexate or csDMARD if rescued) after implementation of Protocol Amendment 6 (December 2019) up to Week 260.
Arm/Group | Weeks 1-24: Methotrexate Monotherapy | Weeks 1-24: Upadacitinib 7.5 mg Monotherapy | Weeks 1-24: Upadacitinib 15 mg Monotherapy | Weeks 1-24: Upadacitinib 30 mg Monotherapy | Weeks 1-260: Methotrexate Monotherapy | Weeks 1-260: Upadacitinib 7.5 mg Monotherapy | Weeks 1-260: Upadacitinib 15 mg Monotherapy | Weeks 1-260/Switch: Upadacitinib 30 mg Monotherapy | Weeks 1-260: Any Upadacitinib 7.5 mg | Weeks 1-260: Any Upadacitinib 15 mg | Weeks 1-260/Switch: Any Upadacitinib 30 mg | After Switch: Upadacitinib 15 mg Monotherapy | After Switch: Any Upadacitinib 15 mg
All-Cause Mortality (participants affected / at risk) | 1/314 | 0/55 | 2/317 | 3/314 | 8/314 | 1/55 | 6/317 | 9/314 | 1/56 | 6/335 | 10/332 | 5/181 | 7/218
Serious Adverse Events (participants affected / at risk) | 13/314 | 5/55 | 16/317 | 20/314 | 49/314 | 13/55 | 68/317 | 71/314 | 15/56 | 88/335 | 79/332 | 28/181 | 35/218
Other Adverse Events (participants affected / at risk) | 159/314 | 38/55 | 169/317 | 174/314 | 234/314 | 52/55 | 242/317 | 256/314 | 55/56 | 272/335 | 277/332 | 100/181 | 126/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 1-24: Methotrexate Monotherapy (N=314) | Weeks 1-24: Upadacitinib 7.5 mg Monotherapy (N=55) | Weeks 1-24: Upadacitinib 15 mg Monotherapy (N=317) | Weeks 1-24: Upadacitinib 30 mg Monotherapy (N=314) | Weeks 1-260: Methotrexate Monotherapy (N=314) | Weeks 1-260: Upadacitinib 7.5 mg Monotherapy (N=55) | Weeks 1-260: Upadacitinib 15 mg Monotherapy (N=317) | Weeks 1-260/Switch: Upadacitinib 30 mg Monotherapy (N=314) | Weeks 1-260: Any Upadacitinib 7.5 mg (N=56) | Weeks 1-260: Any Upadacitinib 15 mg (N=335) | Weeks 1-260/Switch: Any Upadacitinib 30 mg (N=332) | After Switch: Upadacitinib 15 mg Monotherapy (N=181) | After Switch: Any Upadacitinib 15 mg (N=218)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
METABOLIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL FIBROSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHAGIC ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
CATARACT DIABETIC (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MACULAR HOLE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VITREORETINAL TRACTION SYNDROME (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL RECESSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PANCREATIC DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RECTAL POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
GALLBLADDER RUPTURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACTINOMYCOTIC PULMONARY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 3 (3)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 8 (8) | 12 (12)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
CORONAVIRUS PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMALE GENITAL TRACT TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GALLBLADDER ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENITAL HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
HERPES ZOSTER DISSEMINATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTIVE SPONDYLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
KERATITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MENINGITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONEAL TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (2) | 8 (8) | 5 (5) | 1 (2) | 9 (9) | 5 (5) | 1 (1) | 2 (2)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA CRYPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATITIS ESCHERICHIA COLI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Q FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINOBRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL FISTULA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABNORMAL WEIGHT GAIN (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
CENTRAL OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACQUIRED CLAW TOE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBCHONDRAL INSUFFICIENCY FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADENOCARCINOMA GASTRIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGIOFIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG SQUAMOUS CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT PALATE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN GERM CELL TERATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEBACEOUS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE TONGUE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERY DISEASE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MONOPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
MENTAL DISORDER DUE TO A GENERAL MEDICAL CONDITION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RENAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST HYPOPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CERVIX HAEMORRHAGE UTERINE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
EMBOLISM ARTERIAL (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weeks 1-24: Methotrexate Monotherapy (N=314) | Weeks 1-24: Upadacitinib 7.5 mg Monotherapy (N=55) | Weeks 1-24: Upadacitinib 15 mg Monotherapy (N=317) | Weeks 1-24: Upadacitinib 30 mg Monotherapy (N=314) | Weeks 1-260: Methotrexate Monotherapy (N=314) | Weeks 1-260: Upadacitinib 7.5 mg Monotherapy (N=55) | Weeks 1-260: Upadacitinib 15 mg Monotherapy (N=317) | Weeks 1-260/Switch: Upadacitinib 30 mg Monotherapy (N=314) | Weeks 1-260: Any Upadacitinib 7.5 mg (N=56) | Weeks 1-260: Any Upadacitinib 15 mg (N=335) | Weeks 1-260/Switch: Any Upadacitinib 30 mg (N=332) | After Switch: Upadacitinib 15 mg Monotherapy (N=181) | After Switch: Any Upadacitinib 15 mg (N=218)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 6 (8) | 9 (10) | 17 (19) | 4 (4) | 20 (31) | 16 (21) | 5 (5) | 22 (34) | 18 (24) | 4 (4) | 7 (8)
LEUKOPENIA (Blood and lymphatic system disorders) | 4 (5) | 1 (1) | 6 (6) | 4 (4) | 13 (23) | 2 (2) | 9 (19) | 15 (25) | 2 (2) | 11 (24) | 18 (39) | 10 (14) | 10 (14)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 7 (7) | 9 (11) | 11 (15) | 1 (1) | 13 (26) | 25 (37) | 1 (1) | 15 (32) | 27 (56) | 8 (9) | 9 (11)
CATARACT (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (4) | 3 (3) | 2 (3) | 3 (4) | 5 (5) | 3 (4) | 2 (3) | 2 (3)
DRY EYE (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
CHRONIC GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 5 (5) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 13 (13) | 6 (6) | 4 (4) | 12 (13) | 18 (21) | 6 (6) | 13 (14) | 20 (23) | 1 (1) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 4 (5) | 5 (5) | 3 (3) | 4 (5) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 10 (10) | 0 (0) | 11 (12) | 6 (6) | 16 (16) | 3 (3) | 25 (33) | 19 (26) | 3 (3) | 27 (36) | 21 (28) | 3 (3) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 12 (13) | 0 (0) | 8 (8) | 4 (4) | 20 (29) | 1 (1) | 12 (12) | 6 (6) | 1 (1) | 13 (14) | 6 (6) | 1 (1) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 9 (9) | 4 (5) | 7 (7) | 9 (9) | 5 (6) | 8 (8) | 10 (10) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 17 (29) | 1 (2) | 18 (20) | 12 (13) | 29 (47) | 4 (5) | 25 (28) | 17 (19) | 4 (5) | 25 (30) | 19 (22) | 1 (1) | 3 (7)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (2) | 3 (3) | 4 (5) | 8 (10) | 4 (6) | 3 (3) | 8 (10) | 4 (6) | 3 (4) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 7 (8) | 2 (2) | 3 (3) | 1 (1) | 16 (20) | 3 (3) | 1 (1) | 16 (21) | 3 (3) | 1 (1) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 8 (8) | 0 (0) | 7 (8) | 2 (3) | 15 (20) | 1 (1) | 17 (19) | 14 (15) | 1 (1) | 21 (24) | 18 (21) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 6 (6) | 5 (5) | 9 (10) | 9 (9) | 7 (8) | 11 (12) | 9 (9) | 2 (2) | 3 (3)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 6 (6) | 6 (6) | 3 (3) | 8 (8) | 7 (7) | 5 (6) | 5 (6)
BRONCHITIS (Infections and infestations) | 6 (6) | 0 (0) | 7 (8) | 5 (6) | 24 (27) | 7 (9) | 22 (26) | 27 (38) | 9 (11) | 33 (37) | 29 (40) | 5 (9) | 7 (11)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (20) | 4 (4) | 28 (28) | 3 (3) | 4 (4) | 37 (38) | 4 (4) | 19 (20) | 22 (23)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 3 (3) | 7 (7) | 4 (4) | 4 (4) | 9 (9) | 4 (4) | 1 (1) | 1 (1)
CYSTITIS (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 5 (6) | 8 (10) | 9 (9) | 6 (9) | 8 (10) | 11 (11) | 5 (5) | 5 (5)
GASTROENTERITIS (Infections and infestations) | 7 (7) | 2 (2) | 5 (5) | 5 (5) | 12 (12) | 8 (9) | 11 (14) | 10 (11) | 9 (10) | 13 (17) | 10 (11) | 1 (1) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 2 (2) | 7 (8) | 7 (7) | 7 (7) | 12 (12) | 32 (38) | 24 (26) | 13 (13) | 34 (42) | 27 (29) | 7 (8) | 8 (9)
INFLUENZA (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 7 (7) | 8 (8) | 5 (5) | 9 (10) | 10 (10) | 9 (9) | 11 (12) | 2 (2) | 2 (2)
LATENT TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 0 (0) | 11 (11) | 15 (15) | 0 (0) | 14 (14) | 18 (18) | 2 (2) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 13 (15) | 5 (10) | 18 (22) | 17 (18) | 43 (70) | 22 (49) | 48 (87) | 51 (72) | 25 (59) | 57 (99) | 58 (79) | 8 (10) | 10 (12)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (9) | 1 (1) | 4 (5) | 5 (9) | 2 (2) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 8 (10) | 7 (9) | 16 (21) | 11 (13) | 8 (10) | 17 (22) | 13 (16) | 1 (1) | 1 (1)
PERIODONTITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (7) | 4 (4) | 4 (6) | 3 (3) | 5 (5) | 4 (6) | 3 (3) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 6 (6) | 5 (7) | 4 (4) | 8 (9) | 16 (20) | 12 (22) | 12 (14) | 17 (22) | 13 (24) | 14 (18) | 18 (23) | 3 (3) | 4 (4)
SINUSITIS (Infections and infestations) | 6 (6) | 1 (1) | 5 (7) | 4 (4) | 11 (19) | 3 (3) | 14 (27) | 6 (7) | 3 (3) | 16 (29) | 8 (10) | 2 (2) | 3 (3)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 4 (4) | 3 (4) | 3 (3) | 6 (6) | 3 (4) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 (17) | 3 (3) | 20 (23) | 23 (28) | 31 (45) | 9 (14) | 49 (88) | 43 (72) | 9 (14) | 59 (102) | 51 (87) | 5 (7) | 7 (9)
URINARY TRACT INFECTION (Infections and infestations) | 20 (24) | 1 (1) | 17 (19) | 18 (21) | 41 (59) | 1 (3) | 43 (93) | 38 (64) | 1 (3) | 51 (107) | 45 (76) | 13 (14) | 19 (21)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 8 (8) | 8 (10) | 10 (10) | 5 (6) | 10 (12) | 11 (11) | 5 (6) | 3 (4) | 5 (6)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 12 (12) | 2 (2) | 16 (21) | 8 (9) | 28 (34) | 3 (3) | 27 (49) | 28 (48) | 4 (4) | 32 (58) | 32 (52) | 3 (4) | 4 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8 (8) | 0 (0) | 10 (14) | 7 (8) | 23 (27) | 1 (1) | 21 (31) | 24 (33) | 2 (2) | 24 (35) | 27 (36) | 2 (2) | 3 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (3) | 2 (2) | 9 (10) | 34 (39) | 10 (12) | 3 (4) | 37 (68) | 51 (106) | 5 (6) | 46 (79) | 54 (110) | 10 (14) | 12 (17)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 6 (8) | 3 (3) | 6 (10) | 8 (13) | 3 (3) | 9 (14) | 9 (15) | 0 (0) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 3 (3) | 3 (5) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 5 (8) | 3 (4) | 3 (3) | 5 (8) | 4 (5) | 2 (2) | 3 (3)
WEIGHT INCREASED (Investigations) | 2 (2) | 0 (0) | 8 (8) | 2 (2) | 6 (7) | 3 (3) | 15 (17) | 7 (8) | 3 (3) | 17 (19) | 7 (8) | 1 (1) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 5 (7) | 3 (5) | 2 (2) | 7 (9) | 1 (1) | 1 (1)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (6) | 3 (4) | 5 (5) | 15 (17) | 15 (17) | 5 (5) | 17 (22) | 15 (18) | 2 (2) | 2 (2)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 7 (7) | 8 (9) | 2 (2) | 2 (2) | 17 (23) | 14 (19) | 2 (2) | 19 (27) | 16 (21) | 3 (3) | 3 (3)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 2 (2) | 4 (4) | 7 (8) | 6 (6) | 4 (4) | 8 (9) | 8 (9) | 1 (1) | 2 (2)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 11 (12) | 8 (10) | 10 (12) | 0 (0) | 21 (31) | 19 (31) | 0 (0) | 22 (33) | 21 (33) | 4 (4) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 6 (6) | 6 (6) | 13 (14) | 3 (3) | 20 (31) | 16 (19) | 3 (3) | 26 (40) | 17 (22) | 3 (3) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 10 (12) | 6 (7) | 20 (20) | 20 (27) | 6 (7) | 25 (27) | 23 (30) | 6 (6) | 7 (7)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (7) | 1 (1) | 3 (3) | 6 (8) | 1 (1) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 4 (5) | 6 (6) | 3 (3) | 4 (5) | 7 (7) | 5 (5) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 3 (3) | 4 (4) | 8 (8) | 3 (3) | 6 (6) | 8 (8) | 1 (1) | 3 (3)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 19 (20) | 0 (0) | 6 (7) | 1 (1) | 44 (65) | 4 (4) | 29 (37) | 11 (12) | 5 (5) | 39 (57) | 12 (14) | 17 (19) | 25 (31)
DIZZINESS (Nervous system disorders) | 4 (4) | 0 (0) | 5 (5) | 2 (2) | 8 (9) | 4 (4) | 8 (11) | 8 (8) | 4 (4) | 9 (13) | 8 (8) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 6 (6) | 2 (2) | 7 (7) | 14 (16) | 17 (19) | 4 (4) | 12 (13) | 21 (26) | 4 (4) | 18 (20) | 28 (33) | 2 (2) | 4 (4)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (4) | 9 (9) | 1 (1) | 16 (18) | 5 (6) | 2 (2) | 17 (19) | 5 (7) | 1 (1) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 1 (1) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 10 (12) | 10 (11) | 15 (15) | 2 (2) | 24 (28) | 19 (23) | 2 (2) | 29 (35) | 22 (26) | 3 (3) | 3 (3)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 5 (5) | 6 (7) | 6 (7) | 5 (5) | 8 (9) | 6 (7) | 3 (3) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (3) | 5 (6) | 3 (4) | 6 (7) | 5 (6) | 3 (4) | 6 (7) | 5 (6) | 1 (1) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 5 (6) | 4 (4) | 9 (12) | 5 (5) | 8 (9) | 11 (13) | 5 (5) | 9 (10) | 13 (17) | 2 (2) | 2 (2)
HYPERTENSION (Vascular disorders) | 8 (9) | 3 (3) | 12 (12) | 14 (14) | 31 (34) | 8 (9) | 36 (40) | 44 (46) | 9 (10) | 43 (48) | 47 (51) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT02706873/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT02706873/SAP_003.pdf